CLINICAL TRIAL: NCT03729765
Title: A Randomized, Controlled Trial: Hemoperfusion in Extracorporeal Membrane Oxygenation (ECMO) Patients
Brief Title: Hemoperfusion in Extracorporeal Membrane Oxygenation (ECMO) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaotong Hou, Director of Center for Cardiac Intensive Care, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018035X
Record Dates: First submitted 2018-10-30; First posted 2018-11-05 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Cardiogenic Shock
Keywords: veno-arterial extracorporeal membrane oxygenation (VA-ECMO); hemoperfusion; inflammatory factor
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Hemoperfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hemoperfusion (Experimental): The patients in the simultaneous hemoperfusion arm will receive hemoperfusion when extracorporeal membrane oxygenation (ECMO) is commenced. veno-arterial extracorporeal membrane oxygenation (VA-ECMO) patients treat with hemoperfusion three times in a row，each time for 6 hours.
  Interventions: Device: hemoperfusion
- standard care (No Intervention): The patients in the standard care arm will not receive hemoperfusion when lextracorporeal membrane oxygenation (ECMO) is commenced.

INTERVENTIONS:
Device: hemoperfusion — The patients in the simultaneous hemoperfusion arm will receive hemoperfusion when extracorporeal membrane oxygenation (ECMO) is commenced. veno-arterial extracorporeal membrane oxygenation (VA-ECMO) patients treat with hemoperfusion three times in a row，each time for 6 hours.
  Arms: hemoperfusion

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is a temporary mechanical circulatory support device for cardiogenic shock (CS) patients. During extracorporeal membrane oxygenation (ECMO) support, the inflammatory response is intense and complex. It may cause infection, cell damage, organ dysfunction and even death. Hemoperfusion can adsorb inflammatory factors and reduce the inflammatory reaction. CS patients who are likely to receive veno-arterial extracorporeal membrane oxygenation (VA-ECMO) support will be enrolled and randomized with a 1:1 allocation to a simultaneous hemoperfusion arm vs. standard care arm.

1. The patients in the simultaneous hemoperfusion arm will receive hemoperfusion when extracorporeal membrane oxygenation (ECMO) is commenced.
2. The patients in the standard care arm will not receive hemoperfusion when extracorporeal membrane oxygenation (ECMO) is commenced.

The primary outcome is the change of plasma interleukin (IL)-6 level after hemoperfusion is commenced.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years.
2. Admission to ICU.
3. Criteria for the diagnosis of CS as follows: (1) systolic blood pressure less than 90 mmHg for 30 min, a mean arterial pressure less than 65 mmHg for 30 min, or vasopressors required to achieve a blood pressure ≥ 90 mmHg; (2) pulmonary congestion or elevated left-ventricular filling pressures; and (3) signs of impaired organ perfusion with at least one of the following criteria: (a) altered mental status; (b) cold, clammy skin; (c) oliguria; and (d) increased serum lactate.
4. ECMO will supply cardiopulmonary support to the patient
5. The patients will be enrolled and randomized when ECMO is commenced less than 24 hours.

Exclusion Criteria:

1. Refusal of consent.
2. Active hemorrhage or thrombocytopenic purpura
3. BMI≥40
4. Received ECMO bridging to a long-term ventricle assist device or heart transplantation.
5. Infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-19 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
change of plasma interleukin (IL)-6 level | 3 days

SECONDARY OUTCOMES:
change of other inflammatory factor level | 3 days
  plasma interleukin (IL)-1β、8、10（pg/ml）
change of other inflammatory factor level | 3 days
  tumor necrosis factor α (TNF-α)（fmol/ml）
change of other inflammatory factor level | 3 days
  C-reactive protein (CRP)（mg/dl）
All-cause mortality | 30 days
Rate of Multiple organ dysfunction syndrome (MODS) | 30 days
Rate of infection | 30 days
  Any kinds of infection
Duration on extracorporeal membrane oxygenation (ECMO) support | 60 days
Rate of successful weaning from extracorporeal membrane oxygenation (ECMO) | 30 days
  The circulation doesn't deteriorate in 24 hours since weaning from ECMO
Duration on invasive ventilation | 60 days
ICU length of stay | 60 days
Hospital length of stay | 60 days
Rate of adverse event | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dannuo Han, Study Chair — Beijing Anzhen Hospital
Locations (1):
- Center for Cardiac Intensive Care, Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China